CLINICAL TRIAL: NCT00929162
Title: A Phase II, Double-blind, Placebo-controlled, Multi-centre, Randomised Study of ZD4054 (Zibotentan) Plus Carboplatin and Paclitaxel or Placebo Plus Carboplatin and Paclitaxel in Patients With Advanced Ovarian Cancer Sensitive to Platinum-based Chemotherapy
Brief Title: ZD4054 (Zibotentan) or Placebo Plus Chemotherapy in Patients With Advanced Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary objective of the trial was not met and so there was no benefit in collecting further information
Sponsor: AstraZeneca (Industry)
Collaborators: ISTITUTO REGINA ELENA - CENTRO RICERCHE SPERIMENTALI (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4320C00036
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2012-06-06 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Patients With Advanced Ovarian Cancer Sensitive to Platinum-based Chemotherapy
Keywords: ovarian; cancer; chemotherapy; sensitive; ZD4054
MeSH Terms: conditions — Neoplasms; Hypersensitivity | interventions — ZD4054; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZD4054 + paclitaxel + carboplatin (Experimental): ZD4054 10mg oral tablet once daily + paclitaxel +carboplatin intravenous infusions every 3 weeks
  Interventions: Drug: ZD4054 Zibotentan; Drug: Paclitaxel; Drug: Carboplatin
- Placebo + paclitaxel + carboplatin (Placebo Comparator): Placebo oral tablet once daily + paclitaxel +carboplatin intravenous infusions every 3 weeks
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Placebo

INTERVENTIONS:
Drug: ZD4054 Zibotentan — 10 mg oral tablets once daily
  Arms: ZD4054 + paclitaxel + carboplatin
Drug: Paclitaxel — 175mg/m2 IV on day 1 every 3 weeks
Drug: Carboplatin — Carboplatin AUC of 5.0 IV on day 1 every 3 weeks
Drug: Placebo — matching placebo for ZD4054 10 mg
  Arms: Placebo + paclitaxel + carboplatin

SUMMARY:
The purpose of this study is to compare progression-free survival in patients with advanced ovarian cancer treated with ZD4054 in combination with carboplatin+paclitaxel versus placebo in combination with carboplatin+paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of: - Epithelial ovarian carcinoma - Fallopian tube carcinoma - Primary serous peritoneal carcinoma
* Radiologically documented measurable disease according to RECIST criteria assessed by Computerised Tomography (CT) or Magnetic Resonance Imaging MRI) or radiologically documented non-measurable (but evaluable) disease.
* Advanced disease not amenable to curative surgery or radiotherapy at the time of study entry with evidence of disease recurrence or progression at least 6 months following treatment cessation of first-line platinum- containing therapy

Exclusion Criteria:

* Clinical evidence of central nervous system (CNS) metastases
* Non-epithelial ovarian cancer, including malignant mixed Mullerian tumours and mucinous carcinoma of the peritoneum
* Tumour of borderline malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Morris, Study Director — AstraZeneca, Alderley Park; Ian Thomas, Study Chair — AstraZeneca, Alderley Park
Locations (20):
- Germany (13):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Lich
  - Research Site, Magdeburg
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Rostock
  - Research Site, Wiesbaden
- Italy (7):
  - Research Site, Milan, MI
  - Research Site, Perugia, PG
  - Research Site, Aviano, PN
  - Research Site, Roma, Roma
  - Research Site, Campobasso
  - Research Site, Modena
  - Research Site, Napoli

REFERENCES:
- [Derived] Cognetti F, Bagnato A, Colombo N, Savarese A, Scambia G, Sehouli J, Wimberger P, Sorio R, Harter P, Mari E, McIntosh S, Nathan F, Pemberton K, Baumann K. A Phase II, randomized, double-blind study of zibotentan (ZD4054) in combination with carboplatin/paclitaxel versus placebo in combination with carboplatin/paclitaxel in patients with advanced ovarian cancer sensitive to platinum-based chemotherapy (AGO-OVAR 2.14). Gynecol Oncol. 2013 Jul;130(1):31-7. doi: 10.1016/j.ygyno.2012.12.004. Epub 2012 Dec 9. PMID 23234805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 132 patients with advanced ovarian cancer sensitive to platinum-based chemotherapy were recruited between 26th June 2009 and 1st June 2011.
Pre-assignment Details: 12 of the 132 enrolled patients were not randomised to treatment groups as they failed screening
Groups:
- ZD4054+Paclitaxel+Carboplatin: ZD4054 10mg oral tablet once daily + paclitaxel +carboplatin intravenous infusions every 3 weeks
- Placebo+Paclitaxel+Carboplatin: Placebo oral tablet once daily + paclitaxel +carboplatin intravenous infusions every 3 weeks
Period: Overall Study
Arm/Group | ZD4054+Paclitaxel+Carboplatin | Placebo+Paclitaxel+Carboplatin
Started | 59 | 61
Patients Who Received Treatment | 58 | 58
Completed | 11 | 19
Not Completed | 48 | 42
Not completed — Adverse Event | 8 | 5
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol Violation | 32 | 30
Not completed — Other termination reason | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZD4054+Paclitaxel+Carboplatin | Placebo+Paclitaxel+Carboplatin | Total
Number analyzed (Participants) | 59 | 61 | 120
Age Continuous [Mean (Standard Deviation); unit: Years]
  Overall | 57.4 (11.98) | 56.6 (11.07) | 57.0 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 61 | 120
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Median time (in months) from randomisation until clinical progression of disease using the Kaplan-Meier method.
Time Frame: Patients were followed for progression up to 2 years
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054+Paclitaxel+Carboplatin | Placebo+Paclitaxel+Carboplatin
Number analyzed (Participants) | 59 | 61
Months | 7.6 [6.6 to 10.2] | 10.0 [7.1 to 12.2]

2. Secondary Outcome: Overall Survival
Description: Median time (in months) from randomisation until death using the Kaplan-Meier method.
Time Frame: Patients were followed for survival up to 2 years
Population: Overall Survival was not analysed as the study was terminated early.
Arm/Group | ZD4054+Paclitaxel+Carboplatin | Placebo+Paclitaxel+Carboplatin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Tumour Response Rate
Description: Objective response rate defined as participants with a complete or partial response according to RECIST
Time Frame: While receiving paclitaxel + carboplatin study visits were aliged with its administration ie every 3 weeks, then every 6 weeks (up to 2 years)
Population: The number of participants for analysis corresponds to patients with measurable disease at study entry
Measure: Number; unit: Participants
Arm/Group | ZD4054+Paclitaxel+Carboplatin | Placebo+Paclitaxel+Carboplatin
Number analyzed (Participants) | 55 | 58
Participants | 21 | 34

ADVERSE EVENTS:
Arm/Group | ZD4054+Paclitaxel+Carboplatin | Placebo+Paclitaxel+Carboplatin
Serious Adverse Events (participants affected / at risk) | 19/58 | 13/58
Other Adverse Events (participants affected / at risk) | 57/58 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054+Paclitaxel+Carboplatin (N=58) | Placebo+Paclitaxel+Carboplatin (N=58)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 4 | 1
Subileus (Gastrointestinal disorders) | 4 | 0
Ileus (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Toxicity (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
General Physical Health Deterioration (General disorders) | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 5 | 4
Escherichia Infection (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Haemoglobin Decreased (Infections and infestations) | 0 | 1
Ovarian Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Vena Cava Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054+Paclitaxel+Carboplatin (N=58) | Placebo+Paclitaxel+Carboplatin (N=58)
Anaemia (Blood and lymphatic system disorders) | 30 | 25
Neutropenia (Blood and lymphatic system disorders) | 26 | 22
Leukopenia (Blood and lymphatic system disorders) | 20 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 11
Vertigo (Ear and labyrinth disorders) | 2 | 4
Lacrimation Increased (Eye disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 28 | 31
Constipation (Gastrointestinal disorders) | 24 | 19
Vomiting (Gastrointestinal disorders) | 21 | 20
Abdominal Pain (Gastrointestinal disorders) | 16 | 20
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 12
Diarrhoea (Gastrointestinal disorders) | 10 | 12
Stomatitis (Gastrointestinal disorders) | 7 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 4
Fatigue (General disorders) | 20 | 27
Asthenia (General disorders) | 11 | 17
Oedema Peripheral (General disorders) | 13 | 5
Mucosal Inflammation (General disorders) | 9 | 3
Pyrexia (General disorders) | 9 | 7
Oedema (General disorders) | 3 | 0
Drug Hypersensitivity (Immune system disorders) | 15 | 10
Nasopharyngitis (Infections and infestations) | 1 | 9
Influenza (Infections and infestations) | 4 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 6
Bone Pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Headache (Nervous system disorders) | 27 | 17
Paraesthesia (Nervous system disorders) | 11 | 16
Peripheral Sensory Neuropathy (Nervous system disorders) | 10 | 13
Polyneuropathy (Nervous system disorders) | 2 | 9
Dysgeusia (Nervous system disorders) | 4 | 8
Neuropathy Peripheral (Nervous system disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 3 | 5
Depression (Psychiatric disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 10
Dry Skin (Skin and subcutaneous tissue disorders) | 6 | 2
Erythema (Skin and subcutaneous tissue disorders) | 5 | 6
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Hot Flush (Vascular disorders) | 1 | 4
Hypertension (Vascular disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca can review results communications prior to public release and may within 60 days of receipt require amendments to be made. AstraZeneca can also require that submission or disclosure be delayed to allow for the filing of a patent application.